CLINICAL TRIAL: NCT04128930
Title: Ambulatory CPAP Titration in Moderate Obstructive Sleep Apnea
Acronym: ATMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S62965
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed CPAP titration at home (Experimental): Patients will start CPAP treatment with a pressure that is calculated by the following formula (predicted pressure = (0.13 x BMI) + (0.16x neck circumference in cm) + (0.04 x AHI)) with a maximal pressure of 10 cmH2O. After 3 nights and after 7 nights, CPAP data will be remotely evaluated and pressure will be adapted based on the following rules:
  * After 3 nights: median obstructive AHI<5/h: decrease pressure with 2 cmH2O; median obstructive AHI>5/h: increase with 2cmH2O
  * After 7 nights: median obstructive AHI>5/h of 4 nights after last adaptation: increase with 2 cmH2O
  Interventions: Device: PAP titration at home
- APAP titration at home (Active Comparator): Patients will start CPAP treatment with an auto-adjusting CPAP device with pressure levels between 4 and 12 cmH2O. After 7 nights of titration, the optimal pressure will be determined by analyzing the median of the nightly pressure that included 95% of the periods (percentile 95). CPAP treatment will be continued with this fixed optimal pressure.
  Interventions: Device: PAP titration at home

INTERVENTIONS:
Device: PAP titration at home — Fixed CPAP or APAP titration at home

SUMMARY:
The aim of this trial is to compare two different ways of CPAP titration:

CAP titration with fixed pressure vs. auto-titrating CPAP.

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) for the treatment of moderate obstructive sleep apnea (OSA) is only reimbursed in Belgium after in-laboratory overnight titration. Nevertheless, in a recent clinical practice guideline of the AASM, it is recommended that PAP therapy can be initiated using either in-laboratory titration or auto-titrating CPAP (APAP) at home in OSA patients without significant comorbidities. Indeed, several studies evaluated the impact of titration with APAP at home in these patients and showed that the outcome is comparable with in-hospital titration. Up to now, evidence for home titration with fixed CPAP (and follow-up via telemonitoring) is very limited. The use of sleep laboratory space is costly and limits access for diagnostic studies. This study aims to evaluate whether CPAP titration at home with fixed CPAP produces outcomes equal to those following APAP titration.

ELIGIBILITY:
Inclusion Criteria:

* moderate OSA (obstructive AHI 15-30/u on initial PSG)

Exclusion Criteria:

* Presence of hypoventilation
* Presence of central sleep apnea (central AHI ≥ 15)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
CPAP adherence | 3 months
  Usage of the device (mean number of hours/day)

SECONDARY OUTCOMES:
Effective pressure level | 2 weeks
  Optimal pressure of CPAP therapy
Residual apnea/hypopnea index | 2 weeks
  Residual respiratory events during treatment with optimal CPAP pressure during PSG
Mask leaks | 2 weeks
  Objective leaks (L/min) during CPAP treatment
Proportion of good titration | 2 weeks
  Number of patients with residual AHI < 10 (objectivated with PSG)
Residual device AHI | 3 months
  Residual AHI as determined from device data
Epworth Sleepiness Scale | 3 months
  Daytime sleepiness (range: 0-24 - higher score means worse outcome)
Blood pressure | 3 months
  Blood pressure measurement
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  Sleep quality (range: 0-21 - higher score means worse outcome)
36-Item Short Form Health Survey | 3 months
  Quality of life (range: 0-100 - higher score means better outcome)
Hospital contacts | 3 months
  Number of contacts with the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dries Testelmans, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No